CLINICAL TRIAL: NCT02656030
Title: Effects of Specific Training of Deep Cervical Muscles in Chronic Mechanical Neck Pain
Brief Title: Effects of Specific Training for Deep Neck Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thavatchai Suvarnnato, Member of Research Center in Back, Neck, Other Joint Pain and Human Performance, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSuvarnnato
Record Dates: First submitted 2016-01-11; First posted 2016-01-14 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- semispinalis cervicis resisted exercise (Experimental): semispinalis cervicis resisted exercise 2 times/week, 6 weeks duration
  Interventions: Other: semispinalis cervicis resisted exercise
- cranio-cervical flexion exercise (Experimental): cranio-cervical flexion exercise 2 times/week, 6 weeks duration
  Interventions: Other: cranio-cervical flexion exercise
- usual care (Active Comparator): Usual care 2 times/week, 6 weeks duration
  Interventions: Other: usual care

INTERVENTIONS:
Other: semispinalis cervicis resisted exercise — semispinalis cervicis resisted exercise, 2 time per week, 6 weeks duration
  Arms: semispinalis cervicis resisted exercise
Other: cranio-cervical flexion exercise — cranio-cervical flexion exercise, 2 time per week, 6 weeks duration
  Arms: cranio-cervical flexion exercise
Other: usual care — usual care, 2 time per week, 6 weeks duration
  Arms: usual care

SUMMARY:
Recent studies indicate that the patients with chronic neck pain present decreased activation and weak of neck muscles, especially deep flexor and extensor muscles. Alterations of deep are associated with pain and impairment of neck function in chronic neck pain.

Exercise is known to be an important component of treatment programs for patients with neck pain. Recently, many studies have focused on specific training on deep cervical muscles, especially deep cervical flexor and deep cervical extensor muscles.Numerous studies using cranio-cervical flexor exercise as a treatment have revealed reduction on pain, neck disability, changing in activation of deep cervical flexor muscles. Further, the cervical extensor muscles are believed to be equally important for the rehabilitation of patients with neck pain. However, the retention effect of semispinalis cervicis exercise is unknown. Therefore, the semispinalis cervicis exercise still need more evidence to support clinically effects.

The current study will be conducted to fill the gap of the previous study in immediately, short, and long term effects of semispinalis cervicis exercise in chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is a second the most common problems in musculoskeletal problems the low back pain in general population.The prevalence of neck pain at the some point in their lifetime in general population had been reported to be between 43 to 66.7 percent.the neck problems could be involved physical function, psychological function and social function. The economic burden for neck pain is very high.Recent studies indicate that the patients with chronic neck pain present decreased activation and weak of neck muscles, especially deep flexor and extensor muscles. Alterations of deep are associated with pain and impairment of neck function in chronic neck pain.Recently, many studies have focused on specific training on deep cervical muscles, especially deep cervical flexor and deep cervical extensor muscles. The specific training on deep cervical muscles aims to improve control strategy, improve activation of deep cervical flexor muscles to optimize movement control of segmental motion of the cervical spine. Numerous studies using cranio-cervical flexor exercise as a treatment have revealed reduction on pain, neck disability, changing in activation of deep and superficial cervical flexor muscles. Further, the cervical extensor muscles are believed to be equally important for the rehabilitation of patients with neck pain. So, the activation of the deep cervical extensors should be emphasized for the management in people with neck pain. Schomacher et al (2012) suggested that isometric resisted exercise at the second cervical vertebra can improve semispinalis cervicis muscle activity in neck pain patients. However, the retention effect of semispinalis cervicis exercise is unknown. Therefore, the semispinalis cervicis exercise still need more evidence to support clinically effects. The current study will be conducted to fill the gap of the previous study in immediately, short, and long term effects of semispinalis cervicis exercise in chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical neck pain
* Aged between 18 to 59 years
* The symptom more than three months in duration
* A baseline the Thai version of Neck Disability Index (NDI-TH) score of 10 percent or greater

Exclusion Criteria:

* a previous history of whiplash injury
* a previous history injury to the cervical and thoracic spine
* diagnosed with osteoporosis, malignancy or other spinal inflection
* a positive vertebro-basilar artery insufficient test
* diagnosed with cervical radiculopathy and/or myelopathy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | Up to 3-months after the last intervention session

CONTACTS AND LOCATIONS:
Overall Officials: Thavatchai Suvarnnato, M.Sc. PT, Principal Investigator — Research Center in Back, Neck, Other Joint Pain and Human Performance, Khon Kaen University
Locations (1):
- Research Center in Back, Neck, Other Joint Pain and Human Performance, Khon Kaen University, Muang, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Falla D, O'Leary S, Farina D, Jull G. The change in deep cervical flexor activity after training is associated with the degree of pain reduction in patients with chronic neck pain. Clin J Pain. 2012 Sep;28(7):628-34. doi: 10.1097/AJP.0b013e31823e9378. PMID 22156825
- [Result] Schomacher J, Petzke F, Falla D. Localised resistance selectively activates the semispinalis cervicis muscle in patients with neck pain. Man Ther. 2012 Dec;17(6):544-8. doi: 10.1016/j.math.2012.05.012. Epub 2012 Jun 22. PMID 22728210
- [Derived] Suvarnnato T, Puntumetakul R, Uthaikhup S, Boucaut R. Effect of specific deep cervical muscle exercises on functional disability, pain intensity, craniovertebral angle, and neck-muscle strength in chronic mechanical neck pain: a randomized controlled trial. J Pain Res. 2019 Mar 7;12:915-925. doi: 10.2147/JPR.S190125. eCollection 2019. PMID 30881101